CLINICAL TRIAL: NCT03728309
Title: Protocol Title: A Randomized, Multicenter, Evaluator-blind, Controlled Study to Evaluate the Safety and Effectiveness of JUVÉDERM VOLITE™ XC Injectable Gel for the Improvement in Cheek Skin Smoothness
Brief Title: JUVÉDERM® VOLITE™ XC for Cheek Skin Smoothness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1867-701-008
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Skin Smoothness of the Cheeks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- JUVÉDERM® VOLITE™ (Experimental): Participants received an initial treatment of JUVÉDERM® VOLITE™ XC injectable gel, intradermally up to 4 milliliters (mL) on Day 1 followed by an optional touch-up treatment up to 2 mL on Day 30, if applicable. Participants were eligible to receive repeat treatment up to 4 mL at Month 6, if applicable.
  Interventions: Device: JUVÉDERM VOLITE™ XC
- Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ (Experimental): Participants received no treatment for up to 30 days and then received an optional JUVÉDERM® VOLITE™ XC injectable gel initial treatment intradermally up to 4 mLs and an optional touch-up treatment up to 2 mL 30 days later, if applicable.
  Interventions: Device: JUVÉDERM VOLITE™ XC

INTERVENTIONS:
Device: JUVÉDERM VOLITE™ XC — Intradermal, needle in multiple microdepot injections across both cheeks.

SUMMARY:
This is a pivotal study to collect safety and effectiveness data on JUVÉDERM VOLITE™ XC for improvement in skin smoothness of the cheeks in order to support FDA product approval.

ELIGIBILITY:
Inclusion Criteria:

* Ability to follow study instructions and likely to complete all required visits;
* Written informed consent and data privacy consent have been obtained

Exclusion Criteria:

* Has undergone tissue augmentation with dermal fillers including hyaluronic acid (HA), calcium hydroxylapatite, autologous fat, mesotherapy, or other cosmetic procedures (eg, face-lift, laser, photomodulation, intense pulsed light, radiofrequency, dermabrasion, chemical peel, or other ablative procedures) in the fact within 12 months before screening or is planning to undergo any such treatment during the study;
* Has received any crosslinked HA filler in any anatomic area within 12 months of screening;
* Has undergone treatment with botulinum toxin in the cheek area (including crow's feet) within 6 months of screening or is planning to undergo such treatment during the study;
* Has ever received semi-permanent fillers or permanent facial implants (eg, poly-L-lactic acid, polymethylmethacrylate, silicone, expanded polytetrafuoroethylene) anywhere in the face or is planning to be implanted with any of these products at any time during the study;
* Has facial tattoos, piercings, pigmentation, hair (ie, beard, mustache), or past trauma that would interfere with the visualization of the face for the effectiveness assessments;
* Has undergone a dental procedure within 6 weeks before treatment or plans to undergo a dental procedure (other than prophylasix or dental fillings) during the course of the study;
* Has tendency to develop hypertrophic scarring;
* Has a history of allergy to lidocaine, HA products, and/or to gram-positive bacterial proteins as HA is produced by Streptococcus-type bacteria, or is planning to undergo desensitization therapy during the term of the study;
* Has a history of anaphylactic shock;
* Has current cutaneous inflammatory or infectious processes (eg, acne, herpes), abscess, an unhealed wound, or a cancerous or precancerous lesion on the face (injection may be delayed to allow subjects with a history of recurrent oral herpes to take prophylactic antiviral/herpes medication for 2 days);
* Is on an ongoing regimen of anticoagulation therapy (eg, warfarin) or is known to have a coagulation disorder;
* Is on an ongoing regimen of medications (eg, aspirin, ibuprofen) or other substances (eg, herbal supplements with garlic, ginkgo biloba, or ginseng) known to increase coagulation time within 10 days of undergoing study device injection (study device injection may be delayed as necessary to accommodate this 10-day washout period);
* Has active autoimmune disease;
* Has received any investigational product within 30 days before enrollment or is planning to participate in another investigation during the course of this study; - Has begun using any over-the-counter or prescription, oral or topical, anti-wrinkle products on the face within 30 days before enrollment or is planning to begin using such products during the study (subjects who have been on a regimen of such products for at least 30 days are eligible for the study if they intend to continue their regimen throughout the study);
* Females who are pregnant, nursing, or planning a pregnancy during the study;
* Is an employee (or a relative of an employee) of the principal investigator (PI)/evaluating investigator (EI)/treating investigator(TI)/site, Allergan, or representative of Allergan'
* Has a condition or is in a situation which, in the TI's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN, INC., Study Director — Allergan
Locations (14):
- United States (13):
  - Kathleen L. Behr M.D. Inc /ID# 236170, Fresno, California
  - Dermatology Research Associates /ID# 237649, Los Angeles, California
  - Ava MD, Santa Monica, California
  - Art of Skin MD, Solana Beach, California
  - Skin Research Institute LLC, Coral Gables, Florida
  - Advanced Dermatology /ID# 234879, Lincolnshire, Illinois
  - Facial Plastic Surgery Center /ID# 234876, Baltimore, Maryland
  - Skincare Physicians /ID# 235383, Chestnut Hill, Massachusetts
  - Dermatology PartnersInc. /ID# 234946, Wellesley, Massachusetts
  - Dermatology and Laser Surgery Center of New York /ID# 234571, New York, New York
  - Dermatology Laser and Vein Specialists of Carolinas /ID# 236169, Charlotte, North Carolina
  - Clinical Research Center of the Carolinas /ID# 236488, Charleston, South Carolina
  - Dallas Center for Dermatology and Aesthetics /ID# 234452, Dallas, Texas
- Jose Raul Montes Eyes & Facial Rejuvenation, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 209 participants were randomized out of which 202 participants were included in (modified intent-to-treat) mITT population.
Groups:
- JUVÉDERM VOLITE™ XC: Participants received an initial treatment of JUVÉDERM® VOLITE™ XC injectable gel, intradermally up to 4 mL on Day 1 for both cheeks followed by an optional touch-up treatment up to 2 mL on Day 30, if applicable. Participants were eligible to receive repeat treatment up to 4mL at Month 6, if applicable.
Period: Overall Study
Arm/Group | Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ | JUVÉDERM VOLITE™ XC
Started | 73 | 136
mITT Population (mITT Population included all randomized participants who have baseline assessment on the Allergan Cheek Smoothness Scale (ACSS) for both cheeks, and are not in the Fitzpatrick V/VI safety cohort.) | 71 | 131
Volite Treated (VT) Population (VT Population included participants randomized and received VOLITE treatment at the beginning of the Control Period.) | 64 | 135
VOLITE Repeat Treatment (VRT) Population (VRT Population included participants in the VT who received VOLITE repeat treatment.) | 0 | 79
Completed | 61 | 112
Not Completed | 12 | 24
Not completed — Randomized but not Treated | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Lost to Follow-up | 9 | 10
Not completed — Protocol Deviation | 0 | 1
Not completed — Due to COVID | 1 | 3

BASELINE CHARACTERISTICS:
Population: mITT Population included all randomized participants who had baseline assessment on the ACSS scale for both cheeks, and are not in the Fitzpatrick V/VI safety cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ | JUVÉDERM VOLITE™ XC | Total
Number analyzed (Participants) | 71 | 131 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (9.42) | 58.0 (8.24) | 57.1 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 109 | 174
  Male | 6 | 22 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 35 | 56
  Not Hispanic or Latino | 50 | 96 | 146
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 13 | 21
  White | 62 | 115 | 177
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1-point Improvement (Decrease) From Baseline on the Allergan Cheek Smoothness Scale (ACSS) on Both Cheeks at Month 1
Description: The ACSS is a validated 5-point ordinal scale developed by Allergan to grade the severity of skin smoothness on the cheeks. The score ranges from 0 (smooth visual skin texture) to 4 (extremely coarse visual skin texture, crosshatched deep creases, extreme elastosis. Responders are participants with at least 1-point improvement (decrease) from baseline on the ACSS on both cheeks based on evaluating investigator (EI) assessment. Baseline is the last non-missing EI assessment on or before the latter of randomization date or first study treatment date in the control period. The multiple imputation method for the missing data imputation was used for analysis.
Time Frame: Baseline to Month 1
Population: mITT Population included all randomized participants who have baseline assessment on the ACSS scale for both cheeks, and are not in the Fitzpatrick V/VI safety cohort. Missing data in ACSS at Month 1 was imputed using the Multiple Imputation method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ | JUVÉDERM VOLITE™ XC
Number analyzed (Participants) | 71 | 131
percentage of participants | 4.5 [-0.5 to 9.4] | 57.9 [49.3 to 66.6]
Statistical Analysis 1: Comparison: Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ vs JUVÉDERM VOLITE™ XC; Test type: Superiority; p < 0.001, SAS PROC MIANALYZE — The p-value and 95% CI are computed by pooling 30 imputed data sets using SAS PROC MIANALYZE with normal approximation; Percentage Difference = 53.5, 95% CI 2-sided [43.5 to 63.5]

2. Primary Outcome: Number of Participants Who Experience One or More Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical device which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study device. An AE was considered a treatment emergent adverse event (TEAE) if the AE began or worsened (increased in severity or became serious) after first administration of VOLITE for the treatment group and after the date of randomization for the control group.
Time Frame: From first dose of study treatment until 30 days following last dose of study treatment (up to approximately 12 months)
Population: Safety Population included all participants who are randomized and received study intervention (VOLITE or no treatment). A participant was randomized to the JUVÉDERM VOLITE™ XC arm, but not treated in the study. Therefore, this participant was included in the treatment group for the mITT population and in the control group for the safety population
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™: Participants received no treatment for up to 1 month and then received an optional JUVÉDERM® VOLITE™ XC injectable gel initial treatment intradermally up to 4 mLs.
- JUVÉDERM VOLITE™ XC: Participants received an initial treatment of JUVÉDERM® VOLITE™ XC injectable gel, intradermally up to 4 mL on Day 1 followed by an optional touch-up treatment up to 2 mL on Day 30, if applicable. Participants were eligible to receive repeat treatment at Month 6, if applicable.
- Treated Period: VOLITE Post-Control Group: After receiving no treatment in the control period, participants received an initial treatment of JUVÉDERM VOLITE™ XC injectable gel up to 4 mL intradermally followed by an optional touch-up treatment 30 days later, if applicable.
- Repeat Treatment Period: JUVÉDERM® VOLITE™ XC: Participants received an optional repeat treatment of JUVÉDERM® VOLITE™ XC injectable gel, intradermally up to 4 mL at Month 6.
Arm/Group | Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ | JUVÉDERM VOLITE™ XC | Treated Period: VOLITE Post-Control Group | Repeat Treatment Period: JUVÉDERM® VOLITE™ XC
Number analyzed (Participants) | 74 | 135 | 64 | 79
Participants | 5 | 14 | 14 | 5

3. Secondary Outcome: Change From Baseline in Face-Q Satisfaction With Skin Questionnaire at Month 1
Description: The participant assessed satisfaction using the 12 items on the FACE-Q: Satisfaction with Skin questionnaire measured on a 4-point scale where 1=very dissatisfied, 2=somewhat dissatisfied, 3=somewhat satisfied, 4=very satisfied. The responses to the 12 items were summed and converted to a scale score that ranges from 0 (worst) to 100 (best). Higher score indicates more satisfaction. A positive change from baseline indicates improvement.
Time Frame: Baseline and Month 1
Population: mITT Population included all randomized participants who had baseline assessment on the ACSS scale for both cheeks, and are not in the Fitzpatrick V/VI safety cohort. Number analyzed are the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ | JUVÉDERM VOLITE™ XC
Number analyzed (Participants) | 71 | 131
score on a scale
  Baseline | 32.5 (16.53) | 34.3 (17.11)
  Change from Baseline at Month 1: number analyzed (Participants) | 47 | 122
  Change from Baseline at Month 1 | 1.4 (15.18) | 32.0 (27.27)
Statistical Analysis 1: Comparison: Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ vs JUVÉDERM VOLITE™ XC; Test type: Superiority; p < 0.001, 2-sample, t-test; Mean Difference (Final Values) = 28.0, 95% CI 2-sided [21.0 to 36.0], Standard Error of Mean 3.83

4. Secondary Outcome: Percentage of Participants With at Least 1-Point Improvement (Decreased) From Baseline on Both Cheeks in the Allergan Fine Lines Scale (AFLS) Response at Month 1
Description: The AFLS is a validated 5-point ordinal scale developed by Allergan to grade the severity of fine lines on the cheeks. The score ranges from 0 (no fine lines) to 4 (diffuse superficial lines, crosshatching). Responders are participants with at least 1-point improvement (decrease) from baseline on the AFLS on both cheeks based on observed data of EI assessment. Baseline is the last non-missing EI assessment on or before the latter of randomization date or first study treatment date in the control period.
Time Frame: Baseline to Month 1
Population: mITT Population included all randomized participants who had baseline assessment on the ACSS scale for both cheeks, and are not in the Fitzpatrick V/VI safety cohort. Overall number analyzed are the number of participants available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ | JUVÉDERM VOLITE™ XC
Number analyzed (Participants) | 37 | 84
percentage of participants | 5.4 [0.0 to 12.7] | 58.3 [47.8 to 68.9]
Statistical Analysis 1: Comparison: Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ vs JUVÉDERM VOLITE™ XC; Test type: Superiority; p < 0.001, Fisher's Exact Test; Percentage Difference = 52.9, 95% CI 2-sided [40.1 to 65.7] — Comparison of treatment group versus control group at Month 1, responder rate difference, 95% CI for risk difference and p-value was estimated based on Fisher's exact test using mITT population with baseline AFLS score of 2 or 3 on both cheeks

ADVERSE EVENTS:
Time Frame: From first dose of study treatment until 30 days following last dose of study treatment (up to approximately 12 months)
Description: Safety Population: randomized and received intervention (VOLITE or no treatment) as treated. VT Population: randomized and received VOLITE at the start of the Control Period or received optional VOLITE after the Control Period. VRT Population: all in the VT who received VOLITE repeat treatment. A participant was randomized to the JUVÉDERM VOLITE™ XC arm, but not treated. This participant was in the treatment group for the mITT population and in the control group for the safety population.
Groups:
- Treated Period: JUVÉDERM® VOLITE™ XC: Participants received an initial treatment of JUVÉDERM® VOLITE™ XC injectable gel, intradermally up to 4 mL on Day 1 followed by an optional touch-up treatment up to 2 mL on Day 30, if applicable. Participants were eligible to receive repeat treatment at Month 6, if applicable.
Arm/Group | Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ | Treated Period: JUVÉDERM® VOLITE™ XC | Treated Period: VOLITE Post-Control Group | Repeat Treatment Period: JUVÉDERM® VOLITE™ XC
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/135 | 0/64 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/74 | 6/135 | 3/64 | 3/79
Other Adverse Events (participants affected / at risk) | 0/74 | 2/135 | 4/64 | 0/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ (N=74) | Treated Period: JUVÉDERM® VOLITE™ XC (N=135) | Treated Period: VOLITE Post-Control Group (N=64) | Repeat Treatment Period: JUVÉDERM® VOLITE™ XC (N=79)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEMIPLEGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group: No Treatment Then Optional JUVÉDERM® VOLITE™ (N=74) | Treated Period: JUVÉDERM® VOLITE™ XC (N=135) | Treated Period: VOLITE Post-Control Group (N=64) | Repeat Treatment Period: JUVÉDERM® VOLITE™ XC (N=79)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT03728309/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT03728309/SAP_001.pdf